CLINICAL TRIAL: NCT05536505
Title: Adjuvant Treatment Based on Minimal Residual Disease for Resectable Non-squamous Non-Small-Cell-Lung-Cancer With EGFR Mutations
Brief Title: Adjuvant Treatment Based on MRD for EGFR Mutant NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG2105
Record Dates: First submitted 2022-07-21; First posted 2022-09-13 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: MRD
Keywords: NSCLC; Adjuvant; EGFR mutation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRD Positivity Post Operation (Experimental): If MRD confirmed Positivity at either of the two timepoints (Time point 1: blood draw from the 3rd day to 7th day post operation. Time point 2: blood draw on the 28th day post operation), patients would receive icotinib until MRD turned Negativity. During MRD monitoring, icotinib would rechallenge
  Interventions: Genetic: Adjuvant treatment for MRD positivity
- MRD Negativity Post Operation (No Intervention): If MRD confirmed negativity at both of the two timepoints (Time point 1: blood draw from the 3rd day to 7th day post operation. Time point 2: blood draw on the 28th day post operation), patients would receive ctDNA MRD monitoring.

INTERVENTIONS:
Genetic: Adjuvant treatment for MRD positivity — The MRD positive group would receive icotinib as adjuvant treatment. When the peripheral blood MRD turned negative, the subjects entered the drug withdrawal observation period. When the MRD turned positive again, the subjects resumed icotinib treatment. If EGFR T790M mutation was found, researchers would resume medication and choose osimertinib therapy.
  Arms: MRD Positivity Post Operation

SUMMARY:
A prospective, multicenter clinical study designed to explore the efficacy of postoperative adjuvant EGFR-TKIs therapy based on MRD status in patients with stage IB-IIIB EGFR-mutant non-squamous non-small cell lung cancer (non-squamous NSCLC). Primary endpoints include 3-year Disease-Free Survival rate (3y-DFS) and median disease-free survival (mDFS).

DETAILED DESCRIPTION:
All subjects enrolled in this clinical trial will receive peripheral blood MRD status assessment within 1 week and 1 month after surgery, and will be divided into MRD positive group (+) and MRD negative group (-) according to their results , followed by MRD status assessment every 12 weeks.

The MRD positive group would receive icotinib as adjuvant treatment. When the peripheral blood MRD turned negative, the subjects entered the drug withdrawal observation period. When the MRD turned positive again, the subjects resumed icotinib treatment. If EGFR T790M mutation was found, researchers would resume medication and choose osimertinib therapy.

The MRD negative group (-) directly entered the follow-up observation period. When the MRD status of peripheral blood turned positive, the subjects received osimertinib treatment. When the MRD turned negative again, the subjects entered the drug withdrawal observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided.
2. Males or females aged ≥18 years, < 80 years.
3. Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
4. Target population is completely resected pathological stage IB-IIIB NSCLC with EGFR exon 19 deletions, L861Q mutation, G719X mutation and exon 21 L858R activating mutation.
5. Patients who have recovered from R0 resection including lobectomy, sleeve surgery and pneumonectomy.
6. ECOG performance status 0-1.
7. Life expectancy ≥12 weeks.
8. Adequate hematological function: Absolute neutrophil count (ANC) ≥1.8 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
9. Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
10. Adequate renal function: Serum creatinine ≤ 1.25 x ULN, or ≥ 60 ml/min.
11. Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

1. Known severe hypersensitivity to icotinib, osimertinib or any of the excipients of this product.
2. Inability to comply with protocol or study procedures.
3. A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
4. A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease.
5. Interstitial pneumonia.
6. Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, icotinib, cetuximab, trastuzumab).
7. Patients with prior chemotherapy or therapy with systemic anti-tumour therapy (e.g. monoclonal antibody therapy).
8. Patients with prior radiotherapy to primary lesion or lymph nodes.
9. History of another malignancy in the last 5 years with the exception of the following: Other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted. Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
10. Any unstable systemic disease (including active infection, uncontrolled hypertension (systolic pressure > 160mmHg, diastolic pressure > 100mmHg), unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
11. Eye inflammation or eye infection not fully treated or conditions predisposing the subject to this.
12. Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or puts the subject at high risk for treatment-related complications.
13. Patient who has active serious infection (e.g. pyrexia of or 38.0℃ over) Patients who harboring exon 20 T790M mutation, EGFR 20 insertions, ALK fusion, BRAF V600E mutation, MET amplification and KRAS mutation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | From date of opeartion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Disease free survival (DFS)- defined as the time from operation to the first documented disease progression or death, whichever occurs first.
3 yeas DFS rate | From date of opeartion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To compare 3y-DFS rates between the two arms

SECONDARY OUTCOMES:
Overall survival | OS is defined as the time from opeartion to death, regardless of disease recurrence, assessed up to 100 months
  To evaluate the overall survival of both arms

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Chongqing University Three Gorges Hospital, Chongqing
  - The First People's Hospital of Foshan, Foshan
  - Fujian Medical University Union Hospital, Fuzhou
  - Affiliated Cancer Hospital of Guangzhou Medical University, Guangzhou
  - Nanfang Hospital Southern Medical University, Guangzhou
  - Guangdong Provincial People's Hospital, Guanzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of USTC Anhui Provincial Hospital, Hefei
  - The Affiliated Hospital of Inner Mongolia Hospital, Hohhot
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Zhongshan Hospital Fudan University, Shanghai
  - Shenzhen People's Hospital, Shenzhen
  - Tongji Hospital Tongji College of HUST, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zhongshan City People's Hospital, Zhongshan